CLINICAL TRIAL: NCT05560152
Title: Analyzing the Pharmacodynamic Substances and the Effects of Yiqihuayu Decotion for Acute Ischemic Stroke (PHYSIS): A Non-randomized, Controlled Trial
Brief Title: Analyzing the Pharmacodynamic Substances and the Effects of Yiqihuayu Decotion for Acute Ischemic Stroke (PHYSIS)
Acronym: PHYSIS
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ying Gao (Other)
Collaborators: Dongzhimen Hospital, Beijing (Other)
Responsible Party: Sponsor-Investigator, Ying Gao, Professor, Dongzhimen Hospital, Beijing
Organization: Dongzhimen Hospital, Beijing (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2018YFC1705001-05-03
Record Dates: First submitted 2022-09-15; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Ischemic Stroke, Acute
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Experimental: Experimental group Subjects will receive Yiqihuayu Decotion, combined with guidelines-based standard care.
  Interventions:
  Drugs: Yiqihuayu Decotion Other: Standard care (e.g. antiplatelet drugs and statins)
  Interventions: Drug: Yiqihuayu Decotion
- Control group (No Intervention): No Intervention: Control group Subjects will receive guidelines-based standard care.
  Interventions:
  Other: Standard care (e.g. antiplatelet drugs and statins)

INTERVENTIONS:
Drug: Yiqihuayu Decotion — Per os, twice a day, for 7 days.
  Arms: Experimental group

SUMMARY:
The main purposes of this trial are to analyze the pharmacodynamic substances and the effects of Yiqihuayu Decotion for acute ischemic stroke. The trial is a non-randomized, controlled clinical trial.

DETAILED DESCRIPTION:
Yiqihuayu Decotion is effective for acute ischemic stroke clinically, but there is lack of sufficient and reasonable explanation of its intervention effects currently. In order to further clarify the main pharmacodynamic substances of Yiqihuayu Decotion in the treatment of acute ischemic stroke, this study intends to carry out a non-randomized, controlled clinical trial. The primary hypothesis is that, compared with the control group, Yiqihuayu Decotion will produce serial changes in plasma metabolites at pre-dose and 9 days, as well as urine metabolites at pre-dose, 8 days, 9 days and 10 days. The serial changes may be the potential support to explain the intervention effect of Yiqihuayu Decotion. After enrollment, all participants will undergo a 2-day Traditional Chinese Medcine washout period to ensure that the results of pharmacodynamic substances will not be disturbed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Acute ischemic stroke;
* Symptom onset of 4 to 6 days;
* 40 ≤ age ≤ 80 years;
* Be conscious and able to cooperate with clinical information gatherers;
* Patient or legally authorized representative has signed informed consent.

Exclusion Criteria:

* Suspected secondary stroke caused by tumor, brain trauma, or hematological diseases;
* Already dependent in activities of daily living before the present acute stroke (defined as modified Rankin Scale score ≥ 2) ;
* Other conditions that lead to motor dysfunction (e.g., severe osteoarthrosis, rheumatoid arthritis);
* Significant renal or hepatic insufficiency (defined as a serum creatinine concentration, alanine aminotransferase (ALT), or aspartate aminotransferase (AST) value that is twice the upper limit of normal);
* Life expectancy of 3 months or less due to other life-threatening illness (e.g.,advanced cancer)
* Other conditions that render outcomes or follow-up unlikely to be assessed;
* Known to be pregnant or breastfeeding;
* Participating in another clinical study.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09-25 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Differences in Caffeic acid, Amygdalin, Paeoniflorin between experimental group and control group. | 3 days, 8 days, 9 days, 10 days
  Differences in the content of Caffeic acid, Amygdalin, Paeoniflorin in plasma and urine samples between experimental group and control group.

SECONDARY OUTCOMES:
The change of neurological deficits | 1 day, 3 days, 9 days
  The change of neurological deficits is measured by the change of National Institute of Health Stroke Scale (NIHSS) score, ranging from 0 (best score) to 42 (worst score).
The proportion of life dependency | 1 day, 30 days
  The proportion of life dependency is defined as Modified Rankin Scale (mRS) score 0-2. The mRS score ranges from 0 (best score) to 6 (worst score).

IPD SHARING:
Plan to Share IPD: No